CLINICAL TRIAL: NCT06426485
Title: A Multicenter, Randomized Withdrawal, Double-blind, Parallel, Placebo-controlled Design Clinical Trial of Toludesvenlafaxine Hydrochloride Extended-Release Tablets
Brief Title: To Evaluate the Long-term Efficacy and Safety of Toludevenlafaxine Hydrochloride Sustained-release Tablets
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LY03005/CT-CHN-408
Record Dates: First submitted 2024-04-24; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toludesvenlafaxine Hydrochloride Sustained-release Tablets 80 mg or 160 mg group (Experimental): orally once a day
  Interventions: Drug: Toludesvenlafaxine Hydrochloride Sustained-release Tablets
- Placebo (Placebo Comparator): orally once a day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Toludesvenlafaxine Hydrochloride Sustained-release Tablets — orally once a day
  Arms: Toludesvenlafaxine Hydrochloride Sustained-release Tablets 80 mg or 160 mg group
Drug: placebo — orally once a day
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized withdrawal, double-blind, parallel, placebo-controlled design clinical trial of Toludesvenlafaxine Hydrochloride Extended-Release Tablets to evaluate the long-term efficacy and safety in the treatment of Chinese patients with depression.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily signs the informed consent form and is able to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures;
2. Aged 18 years and above, male or female;
3. Outpatients with the main diagnosis of depression meeting DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition) diagnostic criteria for recurrent episodes (without psychotic features) (F33.1/F33.2);
4. MADRS total score ≥ 26 at baseline of screening and open treatment phase.

Exclusion Criteria:

1. Patients who meet the criteria of treatment-resistant depression, that is, patients who have failed to respond to at least two antidepressants with different mechanisms of action in the case of adequate treatment (at least 8 weeks of treatment at the maximum recommended therapeutic dose);
2. Known to have a history of allergy to any component of the investigational product or similar drugs, or allergic constitution (allergic to two or more drugs or food) and the investigator considers it inappropriate to participate in the trial;
3. Significant suicide attempt (defined as a score of ≥ 4 on item 10 of the MADRS scale) or suicidal behavior in the past 6 months on the Columbia-Suicide Severity Rating Scale (C-SSRS) ("actual attempt","interrupted attempt", and"abandoned attempt"with any outcome of"yes");
4. Other diseases meeting DSM-5 diagnostic criteria, including organic mental disorders, substance-related and addictive disorders (except nicotine or caffeine), schizophrenia spectrum and other psychotic disorders, bipolar and related disorders, substance/drug-induced depressive disorders, depressive disorders due to other physical/mental diseases, obsessive-compulsive and related disorders, traumatic and stress-related disorders, dissociative disorders, anorexia nervosa or bulimia, personality disorders;
5. Previous history of increased intraocular pressure or closed glaucoma;
6. Patients with poorly controlled hypertension [screening or baseline sitting systolic blood pressure (SBP) ≥ 160 mmHg or sitting diastolic blood pressure (DBP) ≥ 100 mmHg];
7. Total bilirubin (TBIL) value 1.5 times higher than the upper limit of normal, or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 3 times higher than the upper limit of normal, or creatinine 1.5 times higher than the upper limit of normal at screening;
8. Female patients who are pregnant or have a positive pregnancy test result, or male and female subjects of childbearing potential do not agree to use effective contraception throughout the study and for at least 1 month after discontinuation;
9. Patients who received electroconvulsive therapy (ECT) within 3 months before screening or currently require ECT according to the investigator's judgment;
10. Patients who have received or are receiving systemic psychotherapy (interpersonal therapy, dynamic therapy, cognitive behavioral therapy) within 3 months before screening or currently need systemic psychotherapy according to the investigator's judgment;
11. Patients who received physical therapy such as transcranial magnetic stimulation (TMS), deep brain stimulation, vagus nerve stimulation and transcranial electrical stimulation within 3 months before screening;
12. Patients who received phototherapy within 2 weeks before screening;
13. Patients who have stopped antidepressant drugs for less than 5 half-lives (at least 2 weeks for monoamine oxidase inhibitors (MAOIs) and 1 month for fluoxetine) before enrollment;
14. Those who have participated in other clinical trials within 1 month before screening (excluding those who are not eligible after screening and not enrolled);
15. Currently suffering from acute or severe unstable physical illness, or other conditions that the investigator judges the subject is not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 736 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to relapse. | from Baseline to week 24

SECONDARY OUTCOMES:
Change From Double-Blind Treatment Period Baseline in Montgomery - Eisberg Depression Rating Scale (MADRS) Total Score; | from Baseline to week 24
Change from Double-Blind Treatment Period Baseline in Clinical Global Impression Scale - Severity of Illness (CGI-S) score and Clinical Global Impression Scale - Global Improvement (CGI-I) score | from Baseline to week 24
Change From Double-Blind Treatment Period Baseline in Hamilton Anxiety Rating Scale (HAMA) Total Score. | from Baseline to week 24
Change From Double-Blind Treatment Period Baseline in the Anhedonia Rating Scale (DARS) Score | from Baseline to week 24
Change From Double-Blind Treatment Period Baseline in SHEEHAN Disability Scale (SDS) Score | from Baseline to week 24
Change from Double-Blind Treatment Period Baseline in Digit Symbol Substitution Test (DSST) Score | from Baseline to week 24]

IPD SHARING:
Plan to Share IPD: No